CLINICAL TRIAL: NCT04242069
Title: Healthy for my Baby- A Randomized Controlled Trial Assessing a Preconception Clinically Integrated Technological Intervention to Improve the Lifestyle of Overweight Women and Their Partners
Brief Title: Healthy for my Baby- RCT of a Lifestyle Intervention for Overweight Women in Preconception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-3291
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-12

CONDITIONS: Overweight and Obesity; Pregnancy Complications; Health Behavior; Life Style; Preconception Care
Keywords: Metabolomics
MeSH Terms: conditions — Overweight; Obesity; Pregnancy Complications; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Healthy for my Baby Intervention
  Interventions: Behavioral: Healthy for my Baby
- Control (Other): Usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Healthy for my Baby — Participants will start the preconception intervention by meeting with a health professional for a motivational interview session on healthy lifestyle habits. Following this interview, participants will have access to a mobile phone application that will allow them to track daily lifestyle modification goals. After a month, they will meet the health professional for a second motivational interview and review their progression. Participants will continue to make lifestyle changes through the preconception period by accomplishing smart goals followed daily in the mobile phone application.
  If the woman becomes pregnant, the couple will participate in two more in-person motivational interviews, a month apart. The mobile application will be put in pregnancy mode, and participants will adapt their daily lifestyle goals for the pregnancy. Participants will continue to make lifestyle changes throughout pregnancy by accomplishing smart goals followed daily in the mobile phone application.
  Arms: Intervention
Other: Usual Care — Participants in the control group will receive standard advice on healthy lifestyle habits as provided by their usual care provider. They will receive standard medical care in preconception and pregnancy.
  To improve compliance with the study follow-up, participants in this group will have access to a simplified version of the mobile application that contains a fertility calendar and a research visit calendar. This version of the application does not include lifestyle goals or any information on healthy lifestyle habits.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether an intervention combining motivational interviewing and follow-up with a mobile phone application will help overweight women and their partners adopt healthy lifestyle habits in the preconception period. This study will also evaluate the impact of the intervention on the weight, waist circumference, and body fat of women and their partners. Women and their partners will be followed through pregnancy to explore the effects of the intervention on the adequacy of gestational weight gain, rates of pregnancy complications, delivery mode, and infant birth weight.

DETAILED DESCRIPTION:
In Canada, overweight and obesity are major public health concerns that affect nearly 45% of reproductive-age women. In pregnancy, overweight and excessive gestational weight gain are important risk factors for complications including gestational diabetes, hypertensive disorders of pregnancy, fetal macrosomia, and cesarean delivery. Women who are overweight in pregnancy and who gain excessive weight are also predisposed to subsequent obesity, and their offspring are predisposed to childhood obesity and metabolic syndrome. In light of the failure of pregnancy lifestyle interventions to improve pregnancy outcomes for overweight and obese women, earlier intervention is mandated. Preconception appears as a key period to prevent overweight and pregnancy complications.

The main objective of this study is to evaluate the impact of the Healthy for my Baby intervention on the diet quality of women in the preconception period, as measured with the Canadian Healthy Eating Index 2007 (C-HEI). Urinary profiling of dietary exposure biomarkers will be used as a secondary assessment of diet quality. Secondary outcomes for preconception include the effect of the intervention on the lifestyle habits and anthropometric measures of women and their partners.

In pregnancy, the main secondary objective is to evaluate the impact of the intervention on the pattern of gestational weight gain as defined by the 2009 Institute of Medicine recommendations. Other outcomes for pregnancy include the rates of gestational diabetes, hypertensive disorders of pregnancy, macrosomia, and cesarean delivery. The lifestyle habits of women and their partner and the anthropometric measures of their spouses will also be evaluated in pregnancy. Fertility outcomes will be reported as exploratory measures.

Eligible subjects are couples aged 18 to 40 years who wish to conceive within 12 months of trial inclusion, in which the female partner has a BMI ≥ 25 kg/m2. Exclusion criteria are insufficient knowledge of French or English, an anticipated move to another region, a personal history of infertility, type 1 or 2 diabetes mellitus, prior bariatric surgery, an eating disorder established by clinical diagnosis, medical contraindication to pregnancy, medical contraindication to physical activity, participation in another intensive lifestyle intervention, or a known or anticipated disease or surgery likely to cause an important weight loss. Multiple pregnancies will be excluded from the pregnancy follow-up to limit aberrant data.

Couples will be randomized in blocks to the intervention or control group in a 1:1 ratio with randomly selected block size. The intervention will include two sessions of motivational interviewing on healthy lifestyle in preconception, and two more sessions in pregnancy. As an adjunct to in-person meetings, couples will have access to a mobile phone application to self-monitor daily lifestyle smart goals. Participants in the control group will receive standard advice on lifestyle as provided by their usual care provider. To improve compliance with the study follow-up, participants in this group will have access to a simplified version of the mobile application that contains a fertility calendar and a research visit calendar.

Research visits will take place at study inclusion and every 3 months in preconception for up to 6 months. In pregnancy, study visits will take place in the first (6-8 weeks), second (24-26 weeks), and third (32-34 weeks) trimesters. The C-HEI will be measured at 0, 2, 4, and 6 months in preconception and every trimester in pregnancy with two web-based 24-hour dietary recalls. Urine samples will be collected at 0 and 2 months in preconception and at 24-26 weeks in pregnancy. Data on pregnancy and neonatal outcomes will be collected from medical files at the end of the trial.

A sample size of 54 women is required to detect a 10-point difference in the C-HEI score (maximal value 100) between the groups with an alpha value of 5%, 80% power, and a 13 points standard deviation. Sixty-eight women and their partners will be recruited to account for a 20% attrition rate.

The evolution of the C-HEI score with time in the preconception period will be compared between groups using a mixed linear model. Student's t-test will also be used to compare the average HEI-score between groups at 3, and 6-month follow-up. A statistical significance of 5% with Bonferroni correction for multiple comparisons will be used for the preconception primary outcome assessment. The concentration of 40 urinary metabolites will be compared between baseline, 2 months in preconception and 24-26 weeks of pregnancy using repeated measures ANOVA or Friedman test with a Bonferroni adjustment for multiple comparisons. The proportion of adequate gestational weight gain will be compared between groups with a Chi-squared test. Secondary outcomes will be assessed using Student's t-test, Wilcoxon test, Chi-squared test, or Fisher's exact test as appropriate. For all secondary outcomes statistical significance is set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Women and their partner who wish to conceive within 12 months of trial inclusion
* Woman's body mass index ≥ 25 kg/m2
* Access to a smart phone

Exclusion Criteria:

* Insufficient knowledge of French or English
* Anticipated move to another region
* Personal history of infertility
* Type 1 or 2 diabetes mellitus
* Prior bariatric surgery
* Active eating disorder established by clinical diagnosis
* Medical contraindication to pregnancy
* Medical contraindication to physical activity
* Participation in another intensive lifestyle intervention
* Known or anticipated disease or surgery likely to cause an important weight loss
* Multiple pregnancies will be excluded from the pregnancy follow-up to limit aberrant data

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Women's diet quality in preconception measured with the Canadian-Healthy Eating Index- 2007 | 0, 2, 4, and 6 months
  Women's C-HEI score will be measured with two or three online 24 hour dietary recalls (R24W tool) at each time point. Value range 0-100 with a higher score indicating better diet quality. The change of the score in time during the preconception period will be compared between the groups.

SECONDARY OUTCOMES:
Women's Urinary Food exposure Biomarker Profile | 0 and 2 months in preconception, 24- 26 weeks in pregnancy.
  Three urine spot samples collected over a week will be pooled after normalizing using refractive index measurement to guide dilution. Around 40 metabolites will be targeted for the quantitative measurement of dietary intake biomarker concentrations.
Men and Women's diet quality measured with the Canadian-Healthy Eating Index- 2007. | 0, 2, 4, and 6 months in preconception and 10-12 weeks, 24-26 weeks, and 32-34 weeks in pregnancy.
  The C-HEI score will be measured with two or three online 24 hour dietary recalls at each time point (R24W tool). Value range 0-100 with a higher score indicating better diet quality.
Men and Women's physical activity level measured with the International Physical Activity Questionnaires Short Version. | 0, 3 and 6 months in preconception and 10-12 weeks, 24-26 weeks, and 32-34 weeks in pregnancy.
  Physical activity measured in MET-minutes/week. Value range of 0-5000 MET-minutes/week with a higher score indicating a higher activity level.
Men and Women's steps per day measured with a Fitbit. | 0, 3 and 6 months in preconception and 10-12 weeks, 24-26 weeks, and 32-34 weeks in pregnancy.
  Steps per day measured with a wristband accelerometer over 7 days . Value range 0- 15 000 steps per day with a higher step count indicating a higher activity level.
Men and Women's minutes of moderate and vigorous physical activity measured with a Fitbit. | 0, 3 and 6 months in preconception and 10-12 weeks, 24-26 weeks, and 32-34 weeks in pregnancy.
  Minutes of moderate and vigorous physical activity per week measured with a wristband accelerometer over 7 days. Value range 0-800 minutes with a higher number of minutes indicating a higher activity level.
Men and Women's Sleep quality measured with the Pittsburgh Sleep Quality Index | 0, 3 and 6 months in preconception and 10-12 weeks, 24-26 weeks, and 32-34 weeks in pregnancy.
  Sleep quality measured with a questionnaire. Value range 0-21 with a higher score indicating lower sleep quality.
Men and Women's quality of life measured with the SF-12 v2 | 0, 3 and 6 months in preconception and 10-12 weeks, 24-26 weeks, and 32-34 weeks in pregnancy.
  Quality of life measured with a questionnaire and reported as a t-score. Value range 0-100 with a higher score indicating better quality of life.
Men and Women's Anxiety and Depression symptoms measured with the Hospital Anxiety and Depression Scale. | 0, 3 and 6 months in preconception and 10-12 weeks, 24-26 weeks, and 32-34 weeks in pregnancy.
  Anxiety and Depression symptoms measured with a questionnaire. Value range 0-42 with a higher score indicating more anxiety and depression symptoms.
Women's body fat percentage. | 0, 3, and 6 months in preconception.
  The change in body fat will be assessed in preconception using foot-to-foot bioimpedance.
Women's waist circumference in centimeters. | 0, 3, and 6 months in preconception.
  The change in waist circumference will be assessed in preconception using a measuring tape and a standardized protocol.
Men and Women's weight in kilograms. | 0, 3 and 6 months in preconception and 10-12 weeks, 24-26 weeks, and 32-34 weeks in pregnancy.
  The change in bodyweight will be assessed throughout the study using a calibrated scale.
Men's body fat percentage. | 0, 3 and 6 months in preconception and 10-12 weeks, 24-26 weeks, and 32-34 weeks in pregnancy.
  The change in body fat will be assessed throughout the study using foot-to-foot bioimpedance.
Men's waist circumference in centimeters. | 0, 3 and 6 months in preconception and 10-12 weeks, 24-26 weeks, and 32-34 weeks in pregnancy.
  The change in waist circumference will be assessed throughout the study using a measuring tape and a standardized protocol.
Proportion of adequate gestational weight gain | At delivery.
  Women's total weight gain in pregnancy will be obtained from their medical file. The proportion of adequate gestational weight gain according to BMI specific recommendations (IOM, 2009) will be compared between groups.
Rate of pregnancy complications | At delivery.
  Rates of gestational diabetes (diagnosed with a provoked hyperglycemia test or serial capillary glycemia measures), gestational hypertension (clinical diagnosis), pre-eclampsia (clinical diagnosis), fetal macrosomia (birth weight over the 90th percentile for the gestational age and sex), and mode of delivery.

OTHER OUTCOMES:
Fertility outcomes | After 9 months of follow-up.
  Rates of clinical pregnancies (embryo with a positive heartbeat on first trimester ultrasound), spontaneous miscarriage (unviable pregnancy prior to 20 weeks of gestation), and live birth rate.

CONTACTS AND LOCATIONS:
Overall Officials: William D Fraser, MD,MSc, Principal Investigator — Researcher, Centre de recherche du CHUS
Locations (2):
- Canada (2):
  - Centre de recherche du CHU de Québec Université Laval, Québec, Quebec
  - Centre de recherche du CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Government of Canada SC. Measured adult body mass index (BMI) (World Health Organization classification), by age group and sex, Canada and provinces, Canadian Community Health Survey - Nutrition [Internet]. 2017. Available at: https://www150.statcan.gc.ca/t1/tbl1/en/tv.action?pid=1310079401
- [Background] Marchi J, Berg M, Dencker A, Olander EK, Begley C. Risks associated with obesity in pregnancy, for the mother and baby: a systematic review of reviews. Obes Rev. 2015 Aug;16(8):621-38. doi: 10.1111/obr.12288. Epub 2015 May 28. PMID 26016557
- [Background] Battista MC, Hivert MF, Duval K, Baillargeon JP. Intergenerational cycle of obesity and diabetes: how can we reduce the burdens of these conditions on the health of future generations? Exp Diabetes Res. 2011;2011:596060. doi: 10.1155/2011/596060. Epub 2011 Oct 29. PMID 22110473
- [Background] International Weight Management in Pregnancy (i-WIP) Collaborative Group. Effect of diet and physical activity based interventions in pregnancy on gestational weight gain and pregnancy outcomes: meta-analysis of individual participant data from randomised trials. BMJ. 2017 Jul 19;358:j3119. doi: 10.1136/bmj.j3119. PMID 28724518
- [Background] Institute of Medicine (US) and National Research Council (US) Committee to Reexamine IOM Pregnancy Weight Guidelines; Rasmussen KM, Yaktine AL, editors. Weight Gain During Pregnancy: Reexamining the Guidelines. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK32813/ PMID 20669500
- [Background] Garriguet D. Diet quality in Canada. Health Rep. 2009 Sep;20(3):41-52. PMID 19813438
- [Derived] Hardy I, Lloyd A, Morisset AS, Camirand Lemyre F, Baillargeon JP, Fraser WD. Healthy for My Baby Research Protocol- a Randomized Controlled Trial Assessing a Preconception Intervention to Improve the Lifestyle of Overweight Women and Their Partners. Front Public Health. 2021 Aug 3;9:670304. doi: 10.3389/fpubh.2021.670304. eCollection 2021. PMID 34414154